CLINICAL TRIAL: NCT05760638
Title: Real-World Evidence (RWE) Data Analysis of 1-year Safety, Consistent Utilization, and Consistent Efficacy of Remote Electrical Neuromodulation (REN)
Brief Title: Real-World Evidence (RWE) Data Analysis of 1-year Consecutive Use of Remote Electrical Neuromodulation (REN)
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE004
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-02

CONDITIONS: Migraine
Keywords: Migraine headache; Nerivio; REN
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Nerivio — Remote electrical neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application

SUMMARY:
This is a Post-marketing study investigating the long-term safety, utilization, and efficacy of REN during 12 consecutive months of using Nerivio in migraine patients.

Safety will be assessed by the number and type of adverse events. Utilization will be measured by the number of monthly treatments. Efficacy will be evaluated as a change in headache pain severity and functional disability from baseline to 2 hours post-treatment in at least 50% of the treatments.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, ISRAEL) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients 12 years old and above. It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs, modulated frequency of 100-120 Hz, and up to 40 mA output current which the patient can adjust. The REN device is operated by a designated app that is downloaded to the user's phone prior first use of the Nerivio device.

As part of the sign-up process for the Nerivio app, all patients accept the terms of use which specifies that providing personal information is done on their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback. The app includes a secured, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability (None, Mild limitation, Moderate limitation, Severe limitation), and an indication of which medications, if any, were taken within that 2-hour time window.

Post-marketing surveillance is designed to assess the safety, utilization, and efficacy in larger and more diverse populations and in various real-world environments and situations. As a digital therapeutic device (i.e., electroceutical), the REN device enables prospective collection of electronic patient-reported outcomes in real-world clinical practice.

This post-marketing RWE study investigates the safety and efficacy of the Nerivio treatment by analyzing data of patients who used the Nerivio device for consecutive 12 months (1 year): the following outcome will be assessed:

1. - Safety - all adverse events that were reported within the study's period
2. - Utilization - the number of Nerivio treatments per month
3. - Efficacy - pain relief, freedom from pain, improvement in functional disability, and return to normal function (no disability) at 2 hours post-treatment

Together, these three objectives provide a comprehensive evaluation of long-term safety efficacy in a large real-world dataset

ELIGIBILITY:
Inclusion Criteria:

* Age >12
* REN users across the United States who created Nerivio accounts on October 1st, 2019, and later.
* Had at least one Nerivio treatment per month for 12 consecutive months

Exclusion Criteria:

- Treatments shorter than 30 minutes

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and adolescents (age > 12) who suffers from migraine who are using the Nerivio device for acute treatment of migraine
Sampling Method: Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Device Related Adverse Events | 12 months
  Incidence of device-related adverse events reported by subjects

SECONDARY OUTCOMES:
Long Term Utilization of Nerivio | 12 months
  consistency of monthly usage of Nerivio device during 12 months period
Consistent Headache Relief at 2 Hours Post-treatment | 2 hours
  The proportion of subjects reporting headache relief at 2 hours post-treatment in at least 50% of all their treatments. Headache relief is defined as an improvement from severe or moderate pain to mild or no pain.
  Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain)
Consistent Freedom From Headache at 2 Hours Post-treatment | 2 hours
  The proportion of subjects reporting freedom from headache at 2 hours post-treatment in at least 50% of all their treatments. Pain freedom is defined as the disappearance of headache from severe, moderate, or mild headache at treatment initiation to no headache 2 hours later
  Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain)
Consistent Functional Disability Relief at 2 Hours Post-treatment | 2 hours
  The proportion of subjects who reported having Functional Disability at the beginning of the treatment and reported improvement of at least one level of Functional Disability at 2 hours post-treatment in at least 50% of all their treatments.
  Functional Disability level is reported using a 4-point Likert scale (0-No limitation, 1-Some limitation, 2-Moderate limitation, 3-Severe limitation)
Consistent Functional Disability disappearance at 2 Hours Post-treatment | 2 hours
  The proportion of subjects who reported having Functional Disability at the beginning of the treatment and reported no Functional Disability at 2 hours post-treatment in at least 50% of all their treatments.
  Functional Disability level is reported using a 4-point Likert scale (0-No limitation, 1-Some limitation, 2-Moderate limitation, 3-Severe limitation)

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, PhD, Principal Investigator — Theranica Bio-Electronics Ltd
Locations (2):
- Theranica USA Inc, Bridgewater, New Jersey, United States
- Theranica Bio-Electronics Ltd, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Synowiec A, Stark-Inbar A, Weinstein M, Ironi A, Mauskop A. One-Year Consistent Safety, Utilization, and Efficacy Assessment of Remote Electrical Neuromodulation (REN) for Migraine Treatment. Adv Ther. 2024 Jan;41(1):170-181. doi: 10.1007/s12325-023-02697-6. Epub 2023 Oct 19. PMID 37855973